CLINICAL TRIAL: NCT05340062
Title: The Accuracy of Intracranial Pressure Non Invasive Measurement With Trans Cranial Doppler Versus Invasive Measurement in Pediatric Age
Brief Title: Non Invasive Measurement With Trans Cranial Doppler Versus Invasive Measurement in Pediatric Age
Acronym: nICPped
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, angela amigoni, Medical Doctor, Azienda Ospedaliera di Padova
Other Study IDs: 5210/AO/21
Record Dates: First submitted 2022-03-31; First posted 2022-04-21 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Intracranial Hypertension
Keywords: intracranial hypertension; children; cerebral perfusion
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric patients with ICP device: In children requiring ICP, TCD and ONSD will be measured:
  * within 30 minutes before to the placement of the ICP (if possiblel)
  * at least twice a day after placement of the invasive ICP for the first 48 hours
  Each measurement will include:
  * The measure of the invasive ICP
  * Calculation of invasive CPP (invasive MAP-invasive ICP)
  * TCD: FVs, FVd, FVm, from which the nCPP will be obtained with the formula FVdICP. The nICP will be obtained from invasive MAP minus nCPP.
  * The measurement of the nICP ONSD (2) for a total of 2 measurements preferably from the side where the invasive ICP device is positioned.
  Measurements (TCD and ONSD) will be done by two operators blinded by each other in order to evaluate the inter-operator variability
  Interventions: Device: bedside sonography

INTERVENTIONS:
Device: bedside sonography — TCD and ONSD sonography twice a day per 2 days

SUMMARY:
An increase of intracranial pressure (ICP) is an important cause of secondary brain damage. The gold standard for measuring ICP is represented by invasive positioning of intracranial ICP devices.

The most used non-invasive methods (nICP) are obtained through bed-side ultrasound, routinely used in the management of children in Pediatric Intensive Care: arterial Trancranial Doppler (TCD) and ultrasound measurement of the diameter of the optic nerve sheath (ONSD ).

In this study it is proposed to compare the measurement of nICP obtained by TCD and ONSD versus the measurement obtained by the invasive monitoring (iICP) already present.

DETAILED DESCRIPTION:
An iIncrease in intracranial pressure (ICP) is an important cause of secondary brain damage. The cerebral perfusion pressure (CPP), defined as the mean arterial pressure value (MAP) minus the ICP value (CPP = MAP-ICP), represents the pressure gradient that is responsible for cerebral flow. The gold standard for measuring ICP is represented by invasive methods that are intra-parenchymal or intra-ventricular catheters positions by neurosurgeons. The placement of these catheters can cause complications, mainly bleeding and infections.

The most used non-invasive (nICP) methods are obtained through a medical device such as bed-side ultrasound, routinely used in the management of children in Pediatric Intensive Care: arterial Trancranial Doppler (TCD) and ultrasound measurement of the diameter of the optic nerve sheath (ONSD ).

Arterial TCD is one of the most studied methods in adults for the non-invasive estimation of ICP. Formulas derived from the measurement of cerebral flow velocities (VF) such as the Pulsatility Index (PI) and the formula based on the Diastolic Flow Rate (FVdICP) have been shown to have a correlation with the iICP. According to the literature, a PI> 1 is associated with an ICP value> 20 mmHg. Schmitd, Czosnyka et al. subsequently proposed a new formula for the non-invasive measurement of CPP and therefore of ICP (FVdICP), demonstrating the accuracy of CPP measured with the invasive technique The ONSD is a rapid and repeatable method for making a rapid diagnosis of increased ICP not only in adults but also in children, considering the diameter of the optic nerve sheath equal to 4.5 mm in children as the upper limit of the norm. 1 year of age and 4 mm in children under 1 year.

In this study it is proposed to compare the measurement of nICP obtained with the TCD and with the ONSD versus the measurement obtained by the invasive monitoring (iICP) already present.

ELIGIBILITY:
Inclusion Criteria:

* invasive ICP placement

Exclusion Criteria:

* cranial base fracture
* absent informed consent

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: pediatric patients with planned invasive ICP admitted to PICU
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
comparison between ICP and nICP (measured by TCD) | within 48 hours after the invasive ICP placement
  For each patient with invasive ICP, the nICP (measured by TCD) will be compared. We will collect ICP and nICP in pairs for each measurement ( T1 ) using the same unit of measurement. (During 48 hours we will collect ICP and nICP in pairs 4 times: T1 T2 T3 T4. We will finally evaluate the data in pairs in the total sample).
comparison between ICP and nICP (measured by TCD) | within 48 hours after the invasive ICP placement
  For each patient with invasive ICP, the nICP (measured by TCD) will be compared. We will collect ICP and nICP in pairs for each measurement ( T2 ) using the same unit of measurement. (During 48 hours we will collect ICP and nICP in pairs 4 times: T1 T2 T3 T4. We will finally evaluate the data in pairs in the total sample).
comparison between ICP and nICP (measured by TCD) | within 48 hours after the invasive ICP placement
  For each patient with invasive ICP, the nICP (measured by TCD) will be compared. We will collect ICP and nICP in pairs for each measurement ( T3 ) using the same unit of measurement. (During 48 hours we will collect ICP and nICP in pairs 4 times: T1 T2 T3 T4. We will finally evaluate the data in pairs in the total sample).
comparison between ICP and nICP (measured by TCD) | within 48 hours after the invasive ICP placement
  For each patient with invasive ICP, the nICP (measured by TCD) will be compared. We will collect ICP and nICP in pairs for each measurement ( T4 ) using the same unit of measurement. (During 48 hours we will collect ICP and nICP in pairs 4 times: T1 T2 T3 T4. We will finally evaluate the data in pairs in the total sample).

SECONDARY OUTCOMES:
comparison between ICP and nICP (measured by ONSD) | within 48 hours after the invasive ICP placement
  For each patient with invasive ICP, the nICP (measured by ONSD) will be compared twice a day for 2 days. We will collect ICP and nICP in pairs for each measurement (4 times: T1 T2 T3 T4) using the same unit of measurement and evaluate the data in pairs in the total sample.
interrater reliability for TCD measurement | within 48 hours after the invasive ICP placement
  For each patient with invasive ICP, two nICP measurement by TCD will be performed by two operators blinded each other. We will collect nICP values in pairs (by two operators) for each measurement (2 times) using the same unit of measurement and evaluate the data in pairs in the total sample.
interrater reliability for ONSD measurement | within 48 hours after the invasive ICP placement
  For each patient with invasive ICP, two nICP measurement by ONSD will be performed by two operators blinded each other. We will collect nICP values in pairs (by two operators) for each measurement (2 times) using the same unit of measurement and evaluate the data in pairs in the total sample.

CONTACTS AND LOCATIONS:
Overall Officials: angela amigoni, MD, Principal Investigator — University Hospital of Padova
Locations (6):
- Italy (6):
  - PICU IRCSS Sant'Orsola Malpighi, Bologna
  - PICU Spedali Civili BRescia, Brescia
  - PICU Ospedale Mayer, Florence
  - PICU Ospedale Gaslini, Genova
  - PICU University Hospital Padova, Padua
  - PICU Università Cattolica, Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Czosnyka M, Pickard JD. Monitoring and interpretation of intracranial pressure. J Neurol Neurosurg Psychiatry. 2004 Jun;75(6):813-21. doi: 10.1136/jnnp.2003.033126. PMID 15145991
- [Result] Kochanek PM, Tasker RC, Carney N, Totten AM, Adelson PD, Selden NR, Davis-O'Reilly C, Hart EL, Bell MJ, Bratton SL, Grant GA, Kissoon N, Reuter-Rice KE, Vavilala MS, Wainwright MS. Guidelines for the Management of Pediatric Severe Traumatic Brain Injury, Third Edition: Update of the Brain Trauma Foundation Guidelines, Executive Summary. Neurosurgery. 2019 Jun 1;84(6):1169-1178. doi: 10.1093/neuros/nyz051. PMID 30822776
- [Result] Anderson RC, Kan P, Klimo P, Brockmeyer DL, Walker ML, Kestle JR. Complications of intracranial pressure monitoring in children with head trauma. J Neurosurg. 2004 Aug;101(1 Suppl):53-8. doi: 10.3171/ped.2004.101.2.0053. PMID 16206972
- [Result] Schmidt EA, Czosnyka M, Gooskens I, Piechnik SK, Matta BF, Whitfield PC, Pickard JD. Preliminary experience of the estimation of cerebral perfusion pressure using transcranial Doppler ultrasonography. J Neurol Neurosurg Psychiatry. 2001 Feb;70(2):198-204. doi: 10.1136/jnnp.70.2.198. PMID 11160468
- [Result] Malayeri AA, Bavarian S, Mehdizadeh M. Sonographic evaluation of optic nerve diameter in children with raised intracranial pressure. J Ultrasound Med. 2005 Feb;24(2):143-7. doi: 10.7863/jum.2005.24.2.143. PMID 15661943
- [Result] O'Brien NF, Reuter-Rice K, Wainwright MS, Kaplan SL, Appavu B, Erklauer JC, Ghosh S, Kirschen M, Kozak B, Lidsky K, Lovett ME, Mehollin-Ray AR, Miles DK, Press CA, Simon DW, Tasker RC, LaRovere KL. Practice Recommendations for Transcranial Doppler Ultrasonography in Critically Ill Children in the Pediatric Intensive Care Unit: A Multidisciplinary Expert Consensus Statement. J Pediatr Intensive Care. 2021 Jun;10(2):133-142. doi: 10.1055/s-0040-1715128. Epub 2020 Sep 4. PMID 33884214